CLINICAL TRIAL: NCT01785901
Title: The Asthma Control Rate Achieved by Budesonide/Formoterol in Clinical Practice in China
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-RCN-SYM-2012/1
Record Dates: First submitted 2013-02-05; First posted 2013-02-07 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Asthma
Keywords: asthma; control rate; budesonide/formoterol; Non-Interventional study
MeSH Terms: conditions — Asthma | interventions — Methods

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Target subject population 1500: Asthma patients who have already received the treatment of budesonide/formoterol by physicians' determination and whose medications are aligned with the package insert of budesonide/formoterol approved in China
  Interventions: Other: without interventions

INTERVENTIONS:
Other: without interventions — without interventions

SUMMARY:
This is a multi-centre, cross-sectional study planned to be conducted in China. The study aims to observe about 1500 asthma patients who have already received budesonide/formoterol combination treatment by physicians' determination and whose medications are aligned with the package insert of budesonide/formoterol approved in China.

DETAILED DESCRIPTION:
The asthma control rate achieved by budesonide/formoterol in clinical practice in China.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of asthma at least 6 months;
2. Prescribed with budesonide/formoterol treatment at least 3 months before enrolled;
3. Has used the same maintenance dose of budesonide/formoterol for at least 4 weeks before enrolled.

Exclusion Criteria:

1. Participation in any clinical study within 3 months;
2. Have COPD history/suspicious COPD;
3. ≥ 10 pack years of smoking history
4. Used any other asthma maintenance medication accompanied with budesonide/formoterol within 3 months before enrolled
5. With asthma exacerbation (defined as asthma symptom deterioration resulting oral/rectal/parenteral GCS medication or emergency room treatment or hospitalisation) within 4 weeks before enrolled

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Asthma patients from clinic
Sampling Method: Probability Sample
Enrollment: 1502 (Actual)
Dates: Start 2013-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
The rate of controlled and partly controlled asthma according to the definition of Global Initiative for Asthma | one day

SECONDARY OUTCOMES:
The rate of completely controlled and well controlled asthma according to Asthma Control Test's score | one day
The average frequency of reliever use in previous week | one day

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Research Site, Beijing, Beijing Municipality
  - Research Site, Chongqing, Chongqing Municipality
  - Research Site, Guangzhou, Guangdong
  - Research Site, Harbin, Heilongjiang
  - Research Site, Changsha, Hunan
  - Research Site, Baotou, Inner Mongolia
  - Research Site, Nanjing, Jiangsu
  - Research Site, Qingdao, Shandong
  - Research Site, Chengdu, Sichuan
  - Research site, Hangzhou, Zhejiang
  - Research Site, Wenzhou, Zhejiang

REFERENCES:
- [Background] Makar AB, McMartin KE, Palese M, Tephly TR. Formate assay in body fluids: application in methanol poisoning. Biochem Med. 1975 Jun;13(2):117-26. doi: 10.1016/0006-2944(75)90147-7. No abstract available.
- [Derived] Lin J, Li J, Yu W, Liu Y, Liu C, Chen P, He H, He B, Liu S, Zhou X. A multicenter, cross-sectional, observational study of budesonide/formoterol maintenance and reliever therapy in real-world settings. Respir Med. 2017 Jun;127:45-50. doi: 10.1016/j.rmed.2017.04.004. Epub 2017 Apr 6. PMID 28502418
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1035&filename=NIS-RCN-SYM-2012_1Synopsis.pdf
- See also: Lin et al Asthma Control NIS abstract_2015 APSR. Abstract ID: 310 — http://onlinelibrary.wiley.com/doi/10.1111/resp.12706/epdf